CLINICAL TRIAL: NCT06168955
Title: Study of N-homocysteinylation of Key Proteins in Alzheimer's Disease
Brief Title: Study of N-homocysteinylation of Key Proteins in Alzheimer's Disease (HO-MA)
Acronym: HO-MA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, RENAUD Mathilde, Principal investigator, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2023-A01502-43
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Genetic; N-homocysteinylation
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- alzheimer's disease patients (Experimental): Alzheimer's disease patients with positive biomarkers who started their disease before age 75 and benefited from genetic research.
  Interventions: Other: skin biopsy
- Control group (Other): control cell lines from patients free of alzheimer's disease
  Interventions: Other: skin biopsy

INTERVENTIONS:
Other: skin biopsy — skin biopsy for cell culture and N-homocysteinylation study

SUMMARY:
Alzheimer's disease (AD) is the leading cause of dementia in France. It is a multifactorial pathology, combining genetic and environmental risk factors. Homocysteine, a sulfur-containing amino acid belonging to the methionine-monocarbon cycle, has frequently been found at high levels in neurodegenerative diseases, and in AD in particular. It has been shown on human brain sections that the interaction of homocysteine with tau and MAP1, two key AD proteins, was significantly higher in AD patients than in controls, and corresponded to an N-homocysteinylation type interaction.

This is a prospective study, the main objective of which is to compare MAP1 N-homocysteinylation levels in fibroblasts from individuals with AD versus disease-free cell lines.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* Age of onset of AD < 75 years
* Person with AD with positive CSF biomarkers
* Person who has previously benefited from an analysis of AD genetic characteristics (APP, PSEN1, PSEN2, TREM2, ABCA7, SORL1 genes and ApoE status) and an analysis of monocarbon metabolism genes in the case of biochemical abnormalities by clinical exome, targeted panel or complete exome, and for whom the data set is already available.

Exclusion Criteria:

* Pregnant, parturient or breast-feeding women
* Minor (not emancipated)
* Person of legal age (subject to a legal protection measure)
* Adult unable to give consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
MAP1 homocysteinylation level | Baseline

SECONDARY OUTCOMES:
Homocysteinylation level of tau protein | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde Renaud, Principal Investigator — Central Hospital Nancy
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy, Nancy, France